CLINICAL TRIAL: NCT06810635
Title: Polyphenol Metabotypes in People with Diabetes Type 2
Acronym: PPPIL
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); University of Parma (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0601
Record Dates: First submitted 2024-11-06; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: polyphenol; transit time
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Urine Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool Urine Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- T2DM: persons with type 2 diabetes mellitus
  Interventions: Dietary Supplement: Oral Polyphenol Challenge Test / PPPIL; Diagnostic Test: fasting blood sample; Diagnostic Test: Fasting urine collection; Diagnostic Test: 24 hours urine collection; Other: Questionnaires; Diagnostic Test: Stool collection; Diagnostic Test: Transit time determination
- Non diabetic persons: This cohort is a group without type 2 diabetes or any other chronic illness
  Interventions: Dietary Supplement: Oral Polyphenol Challenge Test / PPPIL; Diagnostic Test: fasting blood sample; Diagnostic Test: Fasting urine collection; Diagnostic Test: 24 hours urine collection; Other: Questionnaires; Diagnostic Test: Stool collection; Diagnostic Test: Transit time determination

INTERVENTIONS:
Dietary Supplement: Oral Polyphenol Challenge Test / PPPIL — Patients will receive a so-called oral polyphenol challenge test. It is a pill containing a multitude of polyphenol classes (doi: 10.1093/cdn/nzac072.020)
Diagnostic Test: fasting blood sample — Fasting blood sample will be obtained for determination of markers of metabolic health.
Diagnostic Test: Fasting urine collection — Subjects collect morning urine (or the urine thereafter ) in a separate urine container and write down the time of urine collection for determination of polyphenol metabolites
Diagnostic Test: 24 hours urine collection — Subjects collect urine over the entire 24h. for determination of polyphenol metabolites
Other: Questionnaires — Questionnaires will be performed to collect information on lifestyle and baseline characteristics: physical activity (IPAQ), sleep (PSQI), drinking and smoking behaviour, drug intake and medical record.
Diagnostic Test: Stool collection — Optional: some subjects collect stool samples to test the capacity of the microbiome to degrade polyphenols with a batch experiment.
Diagnostic Test: Transit time determination — Subjects take a pill containing 90mg of royal blue dye (E133) together with the polyphenol pill to determine their transit time. When their stool discolours, the subjects notify the researcher.

SUMMARY:
This cross-sectional study seeks to characterize the overall polyphenol metabotype in patients with T2DM in comparison to age-matched individuals without diabetes. Additionally, the study aims to identify factors that influence the polyphenol metabotype (transit time and gut microbial capacity to degrade polyphenols in particular).

ELIGIBILITY:
Inclusion Criteria:

* all participants
* between 40-85 years
* age-matched individuals without diabetes
* BMI between 18.5-30
* no metabolic syndrome
* persons with T2DM
* at leats 2 years of clinical diagnoses of T2DM
* stable medication use for at least 1 month

Exclusion Criteria:

* pregnancy of breastfeeding
* in last month
* acute use of anti/pre/probiotics
* start of new drug or dietary supplements
* major changes in diet
* major lifestyle changes
* diseases
* Gastrointestinal diseases (inflammatory bowel disease)
* Bariatric surgery
* Other forms of diabetes (cystic fibrosis/MODY/T1DM)
* Heart problems (NYHA 3/4) or previous cardiovascular events
* Liver problems: non-alcohol steatohepatitis (NASH) and cirrhosis
* Lung problems (COPD - GOLD 3/4), cystic fibrosis
* Uncontrolled thyroid function disruption in the past 6 months
* Intake of coumarin derivatives and direct oral anticoagulant medication
* Anti-cancer treatment: chemo-/immunotherapy
* Immonosuppressants (transplant)
* Antiepileptic drugs

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Flemish T2DM patients and controls from Ghent region.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Differences in polyphenol metabolites in morning urine in persons with type 2 diabetes and in healthy controls. | This will be assessed the morning after ingestion of the pill containing polyphenols
  The study aims to characterize the overall polyphenol metabotype in patients with T2DM compared to age-matched individuals without diabetes. For this purpose we will look at morning urine 24h after ingestion of a polyphenol rich pill.

SECONDARY OUTCOMES:
Differences in polyphenol metabolites in 24h urine in persons with type 2 diabetes and in healthy controls. | Urine will be collected over a 24h period after ingestion of the polyphenol pill.
  For this purpose participants will collect urine over a 24h period
Transit time | baseline
  Along with the ingestion of the polyphenol pill, people will consume E133, a food colorant that will also color the stool.
the capacity of the gut microbiome to degrade polyphenols | baseline
  By using a batch experiment.
Metabolic health | baseline
  This will be determined on the fasting blood samples
lifestyle factors and medical history (A) | baseline
  physical activity, using the validated IPAQ questionnaire
lifestyle factors and medical history (B) | baseline
  Sleep, using the validated PSQI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lapauw, Professor, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All anonymous data will be made available on request after publication also to other researchers.